CLINICAL TRIAL: NCT00005050
Title: A Phase I/II Study of Eniluracil Plus Oral 5-Fluorouracil Combined With Oxaliplatin (FOX-E) in Patients With Previously-Treated Colorectal Cancer
Brief Title: Eniluracil, Fluorouracil, and Oxaliplatin in Treating Patients With Advanced Colorectal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067642; P30CA016087 (NIH); NYU-9907; NCI-G00-1718
Record Dates: First submitted 2000-04-06; First posted 2004-06-08 (Estimated); Last update posted 2011-03-28 (Estimated); Status verified 2011-03

CONDITIONS: Colorectal Cancer
Keywords: stage III colon cancer; stage IV colon cancer; stage III rectal cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — eniluracil; Fluorouracil; Oxaliplatin

INTERVENTIONS:
Drug: ethynyluracil
Drug: fluorouracil
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of combining eniluracil, fluorouracil, and oxaliplatin in treating patients who have advanced colorectal cancer that has been treated previously.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose, dose limiting toxicity, and recommended phase II dose of eniluracil, fluorouracil, and oxaliplatin in patients with previously treated advanced colorectal cancer. II. Determine the response rate in patients treated with this regimen.

OUTLINE: This is a dose escalation study of eniluracil and fluorouracil. Patients receive oral eniluracil and oral fluorouracil twice daily on days 1-21. Patients receive oxaliplatin IV over 2 hours on days 1 and 15. Treatment continues every 4 weeks in the absence of disease progression or unacceptable toxicity. Patients with complete response are treated with 2 more courses and then therapy is stopped. Cohorts of 3-6 patients receive escalating doses of eniluracil and fluorouracil until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose limiting toxicity. The recommended phase II dose (RPTD) is defined as 1 dose level below the MTD. Patients are followed at 1 month.

PROJECTED ACCRUAL: A total of 3-30 patients will be accrued for phase I of the study, and an additional 27-40 patients will be accrued for phase II of the study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed advanced colorectal cancer No more than 2 prior chemotherapy regimens including fluorouracil and/or irinotecan (relapse within 6 months of adjuvant therapy is considered 1 prior regimen) Measurable disease

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-1 Life expectancy: At least 6 months Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL SGOT no greater than 5 times upper limit of normal (ULN) Alkaline phosphatase no greater than 5 times ULN No significant hepatic dysfunction Renal: Creatinine no greater than 1.5 mg/dL Creatinine clearance at least 50 mL/min Cardiovascular: No significant cardiovascular dysfunction Neurologic: No dementia or altered mental status that would preclude informed consent No grade 3 motor or sensory neuropathy No significant neurologic dysfunction Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for 6 months after study No malabsorption syndrome or disease significantly affecting gastrointestinal function that would preclude absorption of eniluracil or fluorouracil No active infection requiring systemic therapy within 1 week of study No known platinum allergy No significant endocrine dysfunction

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics Recovered from prior chemotherapy Endocrine therapy: Not specified Radiotherapy: Recovered from prior radiotherapy Surgery: No major resection of the stomach or proximal small bowel that would preclude absorption of eniluracil or fluorouracil

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-08; Primary Completion 2001-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard S. Hochster, MD, Study Chair — NYU Langone Health
Locations (1):
- Kaplan Cancer Center, New York, New York, United States